CLINICAL TRIAL: NCT03317847
Title: Bromfenac 0.09% Versus Dexamethasone 0.1% Ophthalmic Solutions to Reduce Inflammation After Cataract Surgery
Brief Title: Bromfenac Versus Dexamethasone After Cataract Surgery
Acronym: BVD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Azienda USL Reggio Emilia - IRCCS (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Eudract 2016-004358-14
Record Dates: First submitted 2017-10-19; First posted 2017-10-23 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2019-01

CONDITIONS: Inflammation Eye
MeSH Terms: conditions — Endophthalmitis | interventions — bromfenac; Ophthalmic Solutions; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bromfenac (Experimental): Patients randomized to this arm will receive Bromfenac 0.09 % Ophthalmic Solution BID for 2 weeks
  Interventions: Drug: Bromfenac 0.09 % Ophthalmic Solution
- Dexamethasone (Active Comparator): Patients randomized to this arm will receive Dexamethasone 0.1 % Ophthalmic Suspension QID for one week and BID for the following week
  Interventions: Drug: Dexamethasone 0.1% ophthalmic suspension

INTERVENTIONS:
Drug: Bromfenac 0.09 % Ophthalmic Solution — Patients will self-administer 1 drop of Bromfenac twice daily to the affected eye beginning 1 day after cataract surgery and then continuing through the first 14 days of the postoperative period.
  Other Names: Yellox
  Arms: Bromfenac
Drug: Dexamethasone 0.1% ophthalmic suspension — Patients will self-administer 1 drop of Dexamethasone to the study eye beginning 1 day after cataract surgery 4 times daily during the first postoperative week and 2 times daily in the second postoperative week.
  Arms: Dexamethasone

SUMMARY:
The aim of the study is to compare bromfenac to dexamethasone eye drops to control inflammation after cataract surgery. Inflammation in the anterior chamber of the eye will be measured by a Laser Flare Photometer (LFP).

DETAILED DESCRIPTION:
The BVD study is a phase IV, single centre, randomized, active-control, parallel design, open-label trial comparing Bromfenac ophthalmic solution 0.1% and Dexamethasone ophthalmic suspension 0.1% in patients older than 60 years after unilateral cataract surgery.

A total of 76 patients (38 for each arm) will be included in this study. Patients will be selected among subjects who underwent cataract surgery the day before the study enrolment. Enrolment will take place at the participating hospital.

Eligible subjects will be sequentially assigned, according to a computer-generated randomization list (1:1), to one of the following treatment groups:

* Experimental Arm: Bromfenac ophthalmic solution 0.1% eye drops, 2 times per day in the study eye for two weeks;
* Standard Arm: Dexamethasone ophthalmic suspension 0.1% eye drops, 4 times per day in the study eye for the first week and 2 times per day in the study eye for the second week.

Each group must start the drops the day after cataract surgery, for two weeks.

The first post-operative clinical evaluation is planned the day after cataract surgery. The following procedures will be performed on the study eye and data will be collected during this first clinical encounter:

* Eye Drops Usage training
* Concomitant medications
* Best-corrected Visual Acuity
* Laser Flare Photometry
* Slit lamp biomicroscopy
* Intracular pressure (IOP) with pneumotonometer,
* Dilated fundus ophthalmoscopy
* Ocular Comfort Grading Assessment

At least six post-operative follow-up visits are planned after 3, 7, 9, 11, 14 days (±1 day) and 30 days (±3 days) from cataract extraction plus possible adjunctive controls if problems/complications will occur. The following procedures will be performed on the study eye and data will be collected during all clinical encounters:

* Compliance with study medication
* Concomitant medications
* Best-corrected Visual Acuity (only day 7, 14, 30)
* Laser Flare Photometry
* Optical Coherence Tomography testing (only day 30)
* Slit lamp biomicroscopy (only day 7, 14 and 30)
* IOP with pneumotonometer (only day 7, 14 and 30)
* Dilated fundus ophthalmoscopy (only day 30)
* Ocular Comfort Grading Assessment (only day 7, 14 and 30)
* Adverse events

ELIGIBILITY:
INCLUSION CRITERIA

1. Age > 60 year old.
2. Uneventful cataract surgery. Surgical procedure, as described in the patients chart, should be free of any form of intraoperative complication that may increase postoperative inflammation.
3. Availability of relevant ocular history, including: Best Corrected Visual Acuity testing, Laser Flare Photometry, Optical Coherence Tomography, slit lamp biomicroscopy, intraocular pressure (with pneumotonometer), dilated fundus ophthalmoscopy.
4. Ability and willing to follow all instructions and attend all study visits
5. Ability to self-administer study drug (or have a caregiver available to instill all doses of study drug)
6. Ability and willing to provide informed consent for this study protocol.
7. No ocular, topical, systemic, or inhaled NSAIDs or ocular, topical, or systemic gentamicin, or cyclosporine ophthalmic emulsion within 1 week of investigational product initiation or throughout the duration of the study;
8. No topical, inhaled, or systemic corticosteroids within 15 days or depot corticosteroids within 45 days of the investigational product initiation or or throughout the duration of the study;
9. No oral tamsulosin at any time during the clinical trial;
10. Any ocular, topical, or systemic medication that could interfere with normal lacrimation, wound healing, the investigational product, or the interpretation of clinical trial results.
11. For women, the menopausal state is assumed.

EXCLUSION CRITERIA

1. Ocular exclusion criteria:

   1. history of ocular inflammation or trauma;
   2. history of previous intraocular surgery;
   3. corneal haze, edema or any condition that can interfere with LFP measurement by means of reduced transparency of the cornea;
   4. preoperative LFP value > 12 ph/ms (as per patient' chart)
   5. pseudoexfoliation lentis;
   6. retinal vascular diseases;
   7. diabetic retinopathy;
   8. any variation of the foveal profile at OCT (including macular edema and epiretinal membranes)
   9. moderate to severe forms of age related macular degeneration
   10. presence of any sign of intraocular inflammation (including cells or flare in the anterior chamber) in either eye (including uveitis);
   11. intraoperative complications during the surgical procedure that may increase postoperative inflammation; this includes, in particular, patients with posterior capsule rupture;
   12. marked intraocular inflammation at postoperative day 1, including keratic precipitates or any form of uveitis;
   13. BCVA ≤ 1/10 in the non study eye
2. Systemic exclusion criteria:

   1. inflammatory diseases;
   2. any active or chronic/recurrent disease that was uncontrolled and was likely to affect wound healing;
   3. severe blood dyscrasia or bone marrow suppression;
   4. uncontrolled/unstable peptic ulcer disease
   5. any uncontrolled/unstable pulmonary, cardiac, vascular, autoimmune, hepatic, renal, or central nervous system disease;
3. Known hypersensitivity to bromfenac or to any component of the investigational products, procedural medications, salicylates, or other NSAIDs.
4. Patients cannot be enrolled in another clinical study concurrently

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2017-10-16 (Actual); Primary Completion 2018-06-14 (Actual); Study Completion 2019-12-21 (Actual)

PRIMARY OUTCOMES:
Flare to baseline | Within one month
  Time needed to revert the postoperative flare (measured by laser flare meter in the anterior chamber of the eye) to the preoperative or lower level.
Flare at day 14 | 14 days
  Proportion of patients who will have a postoperative flare at day 14 equal or inferior to the preoperative value in the two groups

SECONDARY OUTCOMES:
Best Corrected Visual Acuity (BCVA) | 14 days
  Proportion of subjects with BCVA equal to 10/10 at day 14 in the two groups
Macular thickness at optical coherence tomography (OCT) | 1 month
  Proportion of patients with central macular thickness greater than 300 microns at day 30 in the two groups
Ocular Comfort Grading Assessment (OCGA) | 14 days
  Safety endpoint: proportion of patients with no ocular discomfort at day 14. Ocular discomfort will be assessed by the OCGA scale. The OCGA measures 7 ocular symptoms (eye pain, tearing, itching, foreign body sensation, photophobia, eye discharge, haziness); at visits, patients will assess the severity by grading each symptom as none (0), mild (1), moderate (2), or severe (3)

CONTACTS AND LOCATIONS:
Overall Officials: Marco Coassin, MD PhD, Principal Investigator — Santa Maria Nuova Hospital IRCCS; Luigi Fontana, Study Chair — Santa Maria Nuova Hospital IRCCS
Locations (1):
- Arcispedale Santa Maria Nuova IRCSS - Ophthalmology, Reggio Emilia, RE, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] De Maria M, Coassin M, Mastrofilippo V, Cimino L, Iannetta D, Fontana L. Persistence of Inflammation After Uncomplicated Cataract Surgery: A 6-Month Laser Flare Photometry Analysis. Adv Ther. 2020 Jul;37(7):3223-3233. doi: 10.1007/s12325-020-01383-1. Epub 2020 May 21. PMID 32440977
- [Derived] Coassin M, De Maria M, Mastrofilippo V, Braglia L, Cimino L, Sartori A, Fontana L. Anterior Chamber Inflammation After Cataract Surgery: A Randomized Clinical Trial Comparing Bromfenac 0.09% to Dexamethasone 0.1. Adv Ther. 2019 Oct;36(10):2712-2722. doi: 10.1007/s12325-019-01076-4. Epub 2019 Sep 3. PMID 31482510